CLINICAL TRIAL: NCT05764707
Title: Assessing Efficacy of Intravenous Acetaminophen for Perioperative Pain Treatment in Spinal Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jingping Wang, MD, Ph.D., Associate Professor of Anaesthesia, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2019P002750
Record Dates: First submitted 2023-02-22; First posted 2023-03-13 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Lumbar; Injury
MeSH Terms: conditions — Wounds and Injuries | interventions — Acetaminophen; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravenous Acetaminophen (Experimental): Intravenous acetaminophen (1000mg) will be administered within 30 minutes of skin closure.
  Interventions: Drug: Acetaminophen
- Intravenous Placebo (Placebo Comparator): Intravenous normal saline will be administered within 30 minutes of skin closure.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetaminophen — Patients will received 1000mg of intravenous acetaminophen within 30 minutes of skin closure.
  Other Names: Tylenol
  Arms: Intravenous Acetaminophen
Drug: Placebo — Patients will received 1000mg of normal saline within 30 minutes of skin closure.
  Other Names: Normal Saline
  Arms: Intravenous Placebo

SUMMARY:
Spinal surgeries are generally associated with intense pain in the postoperative period, especially for the initial few days. The aim of this study is to examine the effect of intraoperative intravenous acetaminophen in spine surgery on postoperative analgesic requirements, pain scores, patient satisfaction, and clinical recovery. Enrolled patients are randomized to receive either intravenous acetaminophen or placebo at the time of surgical closure. It is hypothesized that patients receiving intravenous acetaminophen will have improved pain scores, require less opiate medication, and have better patient satisfaction than those receiving placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing 1-2 levels primary spine surgery ≥18 years old

Exclusion Criteria:

* Chronic opiate users
* More than 3 levels or revision spine surgery
* Liver disease patients include elevated LFT, hepatitis A, hepatitis B or hepatitis C, cirrhosis, fatty liver disease, and any other liver diseases caused by drugs, poisons, or alcohol(s)
* Allergy/hypersensitivity to acetaminophen
* Patients that have used acetaminophen during the 24 hours before their scheduled surgery

Subjects who were unable to communicate in English were further excluded because of their inability to complete the postoperative questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
Worst pain score in the post-anesthesia care unit | Time of postoperative care unit discharge readiness, approximately 3 hours
  The primary outcome will assess worst pain score at the time the patient is ready for post anesthesia care unit discharge using the Revised American Pain Society Patient Outcome Questionnaire. This scale ranges from 0 to 10, with higher values reporting more pain.

SECONDARY OUTCOMES:
Postoperative pain scores | Postoperatively until 72 hours or discharge, approximately three days
  Pain scores will be collected for the first 72 hours or up until discharge, whichever comes first, using clinically documented nursing pain scores. Values will be collected on a scale from 0 to 10 with higher values indicating increased (worst) pain.
Intraoperative opioid consumption | Intraoperatively
  Total cumulative morphine equivalents will be reported while the patient is in the operating room.
Postoperative opioid consumption in the post anesthesia care unit | Postoperatively until time of PACU discharge, approximately 3 hours.
  Total cumulative morphine equivalents will be reported while the patient is in the post anesthesia care unit.
Postoperative opioid consumption after discharge from the postoperative care | Time of discharge from the postoperative care unit until discharge from the hospital, an average of two days
  Total cumulative morphine equivalents will be reported starting from the time the patient is discharged from the post anesthesia care unit until they are discharged from the hospital.
Time to rescue analgesia | Postoperatively until discharge, an average of two days
  The time to rescue analgesia (in minutes) will be assessed.
Patient satisfaction | Time of postoperative care unit discharge readiness, approximately 3 hours.
  Satisfaction with the patient's pain treatment in the hospital will be assessed at the time the patient is ready for discharge from the post anesthesia care unit using the Revised American Pain Society Patient Outcome Questionnaire. This scale ranges from 0 (extremely dissatisfied) to 10 (extremely satisfied).
Length of hospital stay | Postoperatively until discharge, an average of two days
  Length of hospital stay (in days) will be reported.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided